CLINICAL TRIAL: NCT02196363
Title: New Ultrasound Parameters for Predicting Birthweight
Acronym: NUPS
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 10/H1013/9
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Fetal Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant mothers: No intervention

SUMMARY:
Babies that are either very small or very big have increased perinatal morbidity and mortality. Predicting which babies will fall into these groups is traditionally done with risk assessment and third trimester manual palpation, however neither of these techniques are sensitive and a considerable number of affected pregnancies are missed. This results in stillbirth for small babies or birth trauma for larger ones. Serial scanning in the third trimester can improve detection rates but this is expensive and cannot currently be provided to all NHS patients.

A more sensitive test that can be performed earlier in pregnancy would allow identification of at risk pregnancies allowing for increased monitoring. New three dimensional ultrasound techniques that measure volume and volumetric flow have become available that may allow this to happen. This study proposes to trial newer ultrasound techniques on a cohort of pregnant women. The findings from these scans will then be correlated with actual birth weights at the end of pregnancy to determine the ability of these parameters to act as screening tools for babies at the extremes of size.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women the beginning of pregnancy to term

Exclusion Criteria:

* Pregnancies in women previously affected by unclassfied fetal abnormality
* Multiple pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be identified by screening booked scan appointments in regular antenatal clinics. The first approach will be by either the named local investigators
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2010-07; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Kidney volume, thigh volume, placental volume, brain volume, final birthweight | up to 34-36 weeks pregnancy gestation

CONTACTS AND LOCATIONS:
Overall Officials: Ed Johnstone, MBChB PhD MRCOG, Principal Investigator — CMFT
Locations (1):
- Central Manchester University Hospitals NHS Foundation Trust, Manchester, United Kingdom